CLINICAL TRIAL: NCT00950677
Title: The Effect of the Glucagon Suppressors Pramlintide and Exenatide on Postprandial Glucose Metabolism in Children With Type 2 Diabetes Mellitus
Brief Title: The Effect of Byetta and Symlin on Post-meal Meal Blood Sugar Levels in Children With Type 2 Diabetes
Acronym: T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Luisa M. Rodriguez, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-22439; K23DK075931 (NIH)
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; pramlintide; Symlin; exenatide; byetta; glucagon; gastric emptying
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; pramlintide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- exenatide (Active Comparator): exenatide one dose
  Interventions: Drug: Byetta (exenatide)
- pramlintide (Active Comparator): pramlintide one dose
  Interventions: Drug: Symlin (pramlintide)

INTERVENTIONS:
Drug: Byetta (exenatide) — exenatide 5 mcg subcutaneously
  Arms: exenatide
Drug: Symlin (pramlintide) — pramlintide 60 mcg subcutaneously
  Arms: pramlintide

SUMMARY:
The purpose of this study is to see if giving study drugs before a meal may lower blood sugars after the meal. An improvement in blood sugar control may prevent long-term problems of diabetes.

DETAILED DESCRIPTION:
A large study in people with type 2 diabetes (T2DM) showed that lowering blood sugars stopped or delayed the occurrence of health problems. As a result of the study, treatment should try to control blood sugars as near to normal as safely possible.

In people without diabetes, the "after meal" blood sugar level is very carefully controlled by several hormones. Insulin (the hormone that lowers blood sugar) and glucagon (hormone that raises blood sugar) play a key role in keeping this careful balance. Also, we now know of 2 new substances made by the body called amylin and GLP-1 that also help with this careful balance. Amylin is made in the pancreas. GLP-1 is made in the gut. We know that both amylin and GLP-1 are abnormal in people with diabetes.

There are two medicines that may help to control after meal blood sugars from going too high. The medicines are called Symlin (pramlintide) and Byetta (exenatide). Symlin works like amylin. Byetta works like GLP-1. Both medications are very similar in the ways that they work to control blood sugars.

Both medicines help to keep glucagon lower after a meal. They both also help the stomach to digest food more slowly so the blood sugar does not go up too fast after eating. They also help to control how much hunger a person may have before meals. This may help a person to eat less and possibly lose weight. Byetta also seems to help islet cells (cells that make insulin) make more insulin.

Byetta and Symlin are FDA approved for use in adults with T2DM. We want to study these drugs in children with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Children with Type 2 Diabetes,
* Between the ages of 12-21 years,
* Tanner stage 4-5 for pubertal development,
* Menstruating females must have a negative urine pregnancy test for inclusion,
* Must have T2DM for at least 6 months,
* History of negative anti-glutamic acid decarboxylase (GAD) -65 and anti-islet cell antibodies,
* HbA1c < 8.5% and on a stable dose of an oral hypoglycemic agent (with or without insulin) over the last 2 months, or well controlled on diet.

Exclusion Criteria:

* A history of a chronic disease other than diabetes (leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, dyslipidemia, cholelithiasis etc),
* BMI> 40 kg/m2,
* Weight of < 60 kg,
* Female with menstrual irregularities,
* Allergy to local anesthetics (ELAMAX Cream, Ethyl Chloride),
* Evidence or history of chemical abuse,
* Anemia (age specific normal range for hemoglobin will be used),
* Elevated liver enzymes (defined as more than 3 times the upper limit of the normal range for age),
* Elevated BUN or creatinine (defined as more than 3 times the upper limit of the normal range for age),
* Use of medications that may increase the blood sugars and admission to the hospital for diabetes related problems over the last 6 months.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Glucose | 4 hours
  concentration and AUC calculations

SECONDARY OUTCOMES:
glucagon | 4 hrours
  concentration and AUC calculations
gastric emptying | 4 hours
  concentration and AUC calculations
pramlintide concentrations | 4 hours
  concentration and AUC calculations
exenatide concentrations | 4 hours
  concentration and AUC calculations

CONTACTS AND LOCATIONS:
Overall Officials: LUISA M RODRIGUEZ, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No